CLINICAL TRIAL: NCT03375528
Title: Matrix Metalloproteinases Expression in the Neointimal Hyperplasia Induced by Drug Eluting Stent (DES) Implantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dankook University (Other)
Responsible Party: Principal Investigator, Tae Soo Kang, Associate Professor, Dankook University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DankookMMP
Record Dates: First submitted 2017-11-20; First posted 2017-12-18 (Actual); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Coronary Artery Disease; Stent Restenosis
Keywords: Matrix metalloproteinase; neointimal hyperplasia
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ultrasonography, Interventional

STUDY DESIGN:
Intervention Model Description: Patients derived from a population of patients referred to 12 months follow-up coronary angiography for ischemic heart disease who are enable to be performed IVUS will be enrolled in the present trial, between December 2017 and December 2018. The study was an all comers design involving consecutive enrollment of patients with stable angina or acute coronary syndrome who had at least 1 coronary lesion (defined as a stenosis of >50%) suitable for stent implantation 12 months before. The follow-up coronary angiography was performed according to standard techniques by experienced interventionalists only. Instent restenosis was defined as a diameter stenosis ≥50% of the vessel reference diameter by visual assessment. Detailed demographic details including anthropometric measurements, cardiovascular risk factors and medication use were recorded for the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- coronary artery disease patients (Experimental): To define the Matrix metalloproteinases expression level in the neointimal hyperplasia induced by DES implantation
  Interventions: Device: DES implantation

INTERVENTIONS:
Device: DES implantation — Coronary artery intervention using Drug eluting stent and Intravascular Ultrasound is performed.
  Other Names: Intravascular Ultrasound

SUMMARY:
If intimal growth is such that the initial lumen is narrowed significantly, distal blood flow is restricted and chronic tissue ischemia results. This occurs in native coronary arteries and during restenosis after coronary angioplasty or failure of some coronary vein grafts. Stent implantation has become the principal revascularization technique for coronary artery disease. But, in-stent restenosis (ISR) by neointimal hyperplasia persists as a significant limitation of this procedure in the era of drug eluting stent (DES). Coronary intervention might induce an inflammatory response by arterial wall damage, release of inflammatory and chemoattractant factors resulting in leukocyte and platelet activation. Then, Migration and proliferation of neointimal smooth muscle cells together with the deposition of extracellular matrix might lead to the development of ISR.

It is known that matrix metalloproteinases (MMPs) play a key role in the pathogenesis of restenosis by controlling extracellular matrix degradation and the release of matrix-degrading MMPs, including MMP -2 and MMP-9, which facilitate intimal remodeling after angioplasty. Previous studies showed that increased levels of MMPs in coronary arteries undergoing percutaneous intervention may be associated with vascular remodeling and restenosis by promoting migration of vascular smooth muscle cells. Recently, Gregory et al. demonstrated that elevated serum activities of MMP-2 and -9 are associated with dramatically increased restenosis rates after PCI with implantation of DES.

In patients with DESs, determination of MMP levels might be useful for identification of patients who are at high risk for ISR. However, not much is known about the relationship between MMPs and neointimal hyperplasia in patients with DES. In this study, the serum activity of MMP-2 and 9 were investigated in patients who had undergone follow-up coronary angiography with intravascular ultrasound (IVUS), which performed at 9 months post-DES implantation. Our aim was to evaluate if individual or combined levels of MMPs were associated with increased neointimal hyperplasia volume, that is, to evaluate the relationship, correlation between the levels of MMPs and neointimal hyperplasia volume.

DETAILED DESCRIPTION:
Materials and methods Subjects (patients) Patients derived from a population of patients referred to 12 months follow-up coronary angiography for ischemic heart disease who are enable to be performed IVUS will be enrolled in the present trial, between Dec 2017 and Dec 2018. The study was an all comers design involving consecutive enrollment of patients with stable angina or acute coronary syndrome who had at least 1 coronary lesion (defined as a stenosis of >50%) suitable for stent implantation 9 months before. The follow-up coronary angiography was performed according to standard techniques by experienced interventionalists only. In-stent restenosis was defined as a diameter stenosis ≥50% of the vessel reference diameter by visual assessment at the site of the lesion treated with the stent observed in ≥1 multiple projections. The single most severe view was used to categorize the pattern of restenosis as proposed by Mehran et al for classification of in-stent restenotic lesions. Detailed demographic details including anthropometric measurements, cardiovascular risk factors and medication use were recorded for the participants.

Angiographic analysis (QCA-analysis) The off-line quantitative coronary angiographic analysis was performed with an automated edge-detection system (QCA-CMS Version 6.0, Medis, Medical Imaging Systems, Leiden, the Netherlands). The contrast-filled, non-tapered catheter tip was used for calibration. The reference diameter was measured by interpolation. Minimal lumen diameter (before and after PCI) and diameter stenosis (before and after PCI) were measured within the stent and within the 5-mm proximal and distal edges of the stent. Furthermore, we measured vessel size, lesion length, and length of stented segment. All analyses were performed by the same investigator that was blinded to all laboratory results.

IVUS imaging and analysis IVUS imaging was performed after intracoronary administration of 0.2 mg nitroglycerin, using a motorized transducer pullback (0.5 mm/s) and a commercial scanner (Boston Scientific/SCIMED, Minneapolis, MN) consisting of a rotating 40-MHz transducer within a 3.2 Fr imaging sheath. The decision to perform IVUS was at the operator's discretion. All IVUS data were assessed off-line by experienced professionals unaware of the allocated stent type or clinical information. Using computerized planimetry (EchoPlaque 2.7, Indec Systems, Mountain View, CA), stent and reference segments were assessed every 1 mm. In-stent measurements were obtained every 1 mm and included EEM, stent, intra-stent lumen, peristent plaque+media (EEM minus stent), and IH (stent minus intra-stent lumen) areas and volumes. Percent IH was defined as IH divided by stent. All volumes were calculated using the Simpson rule and then normalized by stent length (normalized volume).

Blood samples Blood samples were taken under fasting conditions directly before follow-up angiography. Arterial blood was drawn from the coronary arteries into serum separator tubes and samples serums were allowed to clot for 30 min before centrifugation at 1,000 g for 10 minutes and stored at -70°C until use.

Laboratory measurement Endogenous MMP-2 and MMP-9 were measured in serum using a standardized enzyme-linked immunosorbent assay (ELISA; R&D systems). This system measures the endogenous activity of the specific MMPs.

Sample size estimations:

Sample size calculation was based on the null hypothesis that MMP-2 and/or -9 activity showed no correlation with neointimal hyperplasia volume. Using the Lachin formula, sample size calculations were performed to show the expected correlation coefficient (r) more than 0.40 between both group, two-sided alpha 0.05 and 80% statistical power. Finally, 47 patients were calculated.

Statistical analysis :

Continuous variables are expressed as mean±SD. Categorical variables are summarized as counts and percentages and were compared by the chi-square or by Fisher exact test. Serum levels of MMPs were compared by Student t test or by Mann-Whitney U test. Pearson's correlation was used to correlate MMP levels with neointimal hyperplasia volume. Multiple logistic regression was used to evaluate the interaction between variables and MMPs in correlation with neointimal hyperplasia volume and in-stent restenosis. A stepwise entry procedure was applied to identify significant or suggestive (p < 0.1) confounders of either patient group or MMP level. Odds ratios were expressed with 95% confidence intervals. A p-value of less than 0.05 was considered statistically significant. All statistical analyses were performed with the statistical software package SPSS version 12.0 (SPSS, Inc., Chicago, Illinois). The authors had full access to the data and take responsibility for its integrity. All authors have read and agree to the manuscript as written.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic heart disease

Exclusion Criteria:

* Left main coronary artery disease (defined as a stenosis of > 50%)
* Prior complex lesion morphologies (aorto-ostial, bifurcation with >2.0 mm side branch, severe calcification, chronic total occlusion)
* Long lesion that require more than two stents
* Inflammatory conditions likely to be associated with an acute phase response, autoimmune and neoplastic disease
* Advanced liver disease, renal failure, and valvular heart disease
* If there was persistent cardiogenic shock, refractory pulmonary edema, or hemodynamic instability (blood pressure <90/50 mmHg).

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
Matrix Metalloproteinase expression correlate with neointimal plaque volume measure by intravascular ultrasound at 12 months follow up coronary angiography | One time frame - MMP sampling at 12 month follow up coronary angiography.
  Endogenous MMP-2 and MMP-9 were measured in serum using a standardized enzyme-linked immunosorbent assay (ELISA; R&D systems). This system measures the endogenous activity of the specific MMPs. Neointimal plaque volume measure by intravascular ultrasound at 12 months follow up coronary angiography

CONTACTS AND LOCATIONS:
Overall Officials: Tae Soo Kang, PhD, Principal Investigator — Dankook University Hospital 201 Manghyanro, Dongnam-gu, Cheonan-si, Chunchungnam-do, 31116, Republic of Korea

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 1 year of study completion.
Access Criteria: Data acess requests will be reviewed by an external independent Review Panel.

REFERENCES:
- [Background] Katsaros KM, Kastl SP, Zorn G, Maurer G, Wojta J, Huber K, Christ G, Speidl WS. Increased restenosis rate after implantation of drug-eluting stents in patients with elevated serum activity of matrix metalloproteinase-2 and -9. JACC Cardiovasc Interv. 2010 Jan;3(1):90-7. doi: 10.1016/j.jcin.2009.10.023. PMID 20129576
- [Background] Schoenhagen P, Vince DG, Ziada KM, Kapadia SR, Lauer MA, Crowe TD, Nissen SE, Tuzcu EM. Relation of matrix-metalloproteinase 3 found in coronary lesion samples retrieved by directional coronary atherectomy to intravascular ultrasound observations on coronary remodeling. Am J Cardiol. 2002 Jun 15;89(12):1354-9. doi: 10.1016/s0002-9149(02)02346-9. PMID 12062727